CLINICAL TRIAL: NCT03400098
Title: Expanded Access Program for Inotersen (ISIS 420915) in Patients With Hereditary Transthyretin Amyloidosis (hATTR)
Brief Title: ATTR Expanded Access Program (EAP) by Ionis
Status: Approved for marketing | Type: Expanded Access
Sponsor: Ionis Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: ISIS 420915-CS5
Record Dates: First submitted 2018-01-08; First posted 2018-01-17 (Actual); Last update posted 2019-08-05 (Actual); Status verified 2019-08

CONDITIONS: Amyloidosis, Hereditary
MeSH Terms: conditions — Amyloidosis, Familial | interventions — Inotersen

STUDY DESIGN:
Expanded Access Types: Treatment

INTERVENTIONS:
Drug: Inotersen — Inotersen administered by subcutaneous (SC) injections in the abdomen, thigh, or upper arm

SUMMARY:
The purpose of this program is to provide expanded access to Inotersen for up to 100 Patients with Hereditary Transthyretin Amyloidosis (hTTR).

DETAILED DESCRIPTION:
The Program is intended to provided expanded access to Inotersen for eligible patients with hATTR who have limited or no available treatment options.

ELIGIBILITY:
Inclusion Criteria:

* Male or female at least 18 years of age with a diagnosis of hATTR
* Symptoms consistent with polyneuropathy
* Meet Polyneuropathy Disability (PND) Stage I-III requirements

Exclusion Criteria:

* Known Primary Amyloidosis, Leptomeningeal Amyloidosis or Monoclonal Gammopathy of Undetermined Significance or Multiple Myeloma
* Have inadequate cardiac function
* Have low platelet counts
* Have inadequate renal function

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult